CLINICAL TRIAL: NCT02180828
Title: An Case-controlled Randomized Study to the Efficacy of Clotrimazole Vaginal Tablet vs Fluconazole for Severe Vulvovaginal Candidiasis
Brief Title: Clotrimazole Vaginal Tablet vs Fluconazole for Severe Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Shenzhen Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Shangrong Fan, Prof of Dept of Obstetrics and Gynecology, Peking University Shenzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pkuszh-2014-02
Record Dates: First submitted 2014-06-30; First posted 2014-07-03 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Candidiasis, Vulvovaginal
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clotrimazole vaginal tablet (Experimental): 2 doses of 500 mg Clotrimazole administered intravaginally (at day1 and day4)
  Interventions: Drug: Clotrimazole vaginal tablet
- Fluconazole (Active Comparator): 2 doses of 150 mg oral Fluconazole (at day1 and day4)
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Clotrimazole vaginal tablet — 2 doses of 500 mg Clotrimazole administered intravaginally (at day1 and day4)
  Other Names: Canesten
  Arms: Clotrimazole vaginal tablet
Drug: Fluconazole — 2 doses of 150 mg oral Fluconazole (at day1 and day4)
  Other Names: Diflucan
  Arms: Fluconazole

SUMMARY:
The study is focused to prove that the efficacy and safety of Clotrimazole vaginal tablet vs Fluconazole for the treatment of severe vulvovaginal candidiasis

DETAILED DESCRIPTION:
The current study is evaluating both the efficacy and safety of the 2 doses of 500 mg clotrimazole vaginal tablet administered intravaginally( at day 1 and day 4) v.s 2 doses of 150 mg fluconazole( at day 1 and day 4) for treatment of severe vulvovaginal candidiasis.The number of participants with adverse events as a measure of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Vulvovaginal candidiasis infection is diagnosed, the symptoms evaluated using a numerical rating system based on severity (absent=0; mild=1; moderate=2; severe=3) with a minimum VVC Composite Signs/Symptoms score of 7
2. Subject completes the informed consent process
3. Subject agrees to take study medication when scheduled
4. Subject complies with all clinical trial instructions. Commits to all follow-up visits

Exclusion Criteria:

1. had any other sexually transmitted disease or gynaecological abnormality requiring treatment
2. had a disease known to predispose to candidiasis such as diabetes mellitus, or were receiving antibiotics or corticosteriods
3. were pregnant
4. had used antifungal medication in the week before entry
5. were expected to menstruate within seven days of the start of treatment
6. infected more than one candida species

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shangrong Fan, M.D., Principal Investigator — Peking University Shenzhen Hospital
Locations (1):
- Peking University Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
http://onlinelibrary.wiley.com/doi/10.1111/myc.12485/epdf

REFERENCES:
- [Result] Zhou X, Li T, Fan S, Zhu Y, Liu X, Guo X, Liang Y. The efficacy and safety of clotrimazole vaginal tablet vs. oral fluconazole in treating severe vulvovaginal candidiasis. Mycoses. 2016 Jul;59(7):419-28. doi: 10.1111/myc.12485. Epub 2016 Apr 13. PMID 27073145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Started | 120 | 120
Completed | 115 | 113
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 120 | 120 | 240
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6) | 29 (7) | 29 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 120 | 240
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Efficacy 1
Description: The clinical cure rates of clotrimazole and fluconazol: Clinical cure was defined as the resolution of symptoms present at baseline with a total severity score of ≤2. Improvement was defined as considerable reduction in the severity of baseline signs and symptoms with a decrease in the total score by ≥50%.Patients not clinically cured or showing improvement were considered clinical failures.
Time Frame: 7-14 days after treatment (=visit 2)
Population: PPS
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 114 | 110
participants | 102 | 98
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Non-Inferiority or Equivalence — Yes; p = 0.925, Chi-squared

2. Primary Outcome: Therapeutic Efficacy 2
Description: The clinical cure rates of clotrimazole and fluconazol
Time Frame: at days 30-35 follow-up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 114 | 109
participants | 82 | 85
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Non-Inferiority or Equivalence — Yes; p = 0.298, Chi-squared

3. Primary Outcome: Therapeutic Efficacy 3
Description: Mycological cure of clotrimazole group and fluconazole group
Time Frame: at days 7-14 follow-up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 115 | 110
participants | 90 | 81
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Non-Inferiority or Equivalence — 90% power and a two-sided alpha level of 0.05; p = 0.147, Chi-squared

4. Primary Outcome: Therapeutic Efficacy 4
Description: Mycological cure of clotrimazole group and fluconazole group: Mycological cure or failure was referred to as Candida negative or positive,respectively, on Candida culture at follow-up visits.
Time Frame: at days30-35 follow-up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 114 | 109
participants | 62 | 61
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Non-Inferiority or Equivalence — Yes; p = 0.147, Chi-squared

5. Secondary Outcome: Adverse Events 1
Description: Systemic: weak, palpitation, tachycardia, migraine, headache, dizzy, rhinorrhea, numb, dizziness, fatigue.
Time Frame: at day 7-14 follow up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 115 | 113
participants | 1 | 9
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Superiority or Other; p = 0.010, Chi-squared

6. Secondary Outcome: Adverse Events 2
Description: Vulvovaginal pruritus, burning, irritation, and bleeding
Time Frame: at day 7-14 follow up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 115 | 113
participants | 12 | 1
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Superiority or Other; p = 0.002, Chi-squared

7. Secondary Outcome: Adverse Events 3
Description: Gastrointestinal tract: abdominal pain, diarrhoea, nausea
Time Frame: at day 7-14 follow up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 115 | 113
participants | 3 | 3
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Superiority or Other; p = 0.658, Chi-squared

8. Secondary Outcome: Adverse Events 4
Description: Skin sensitivity, urticaria rash, erythematous rash, irritation
Time Frame: at day 7-14 follow up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 115 | 113
participants | 0 | 3
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Superiority or Other; p = 0.123, Chi-squared

9. Secondary Outcome: Total Adverse Events
Description: Total adverse events(cases)
Time Frame: at day 7-14 follow up
Measure: Number; unit: participants
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Number analyzed (Participants) | 115 | 113
participants | 16 | 12
Statistical Analysis 1: Comparison: Clotrimazole Vaginal Tablet vs Fluconazole; Test type: Superiority or Other; p = 0.274, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 month
Description: The adverse events of clotrimazole vaginal tablet were mainly local and mild. Most of the adverse events of fluconazole were systemic.
Arm/Group | Clotrimazole Vaginal Tablet | Fluconazole
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/113
Other Adverse Events (participants affected / at risk) | 13/115 | 10/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clotrimazole Vaginal Tablet (N=115) | Fluconazole (N=113)
Systemic (Cardiac disorders) | 1 (1) | 9 (9) — Systemic: weak, palpitation, tachycardia, migraine,headache, dizzy, rhinorrhea, numb, dizziness, fatigue.
Vulvovaginal (Reproductive system and breast disorders) | 12 (12) | 1 (1) — Vulvovaginal pruritus, burning, irritation, and bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No